CLINICAL TRIAL: NCT05777980
Title: Evaluating the Nutrition Status and Oral Health Impact Profile (OHIP) in Fully Edentulous Patients After Implant-supported Overdenture Rehabilitation: A Prospective Observational Follow-up Study
Brief Title: Effect of Prosthetic Rehabilitation on Nutritional Status of Geriatric Patients
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Ferit Bayram, Assist Prof., Marmara University
Other Study IDs: MU_DHF_SBF_04
Record Dates: First submitted 2023-02-16; First posted 2023-03-21 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Nutrition Disorders; Edentulous Jaw
Keywords: Aged Nutrition Physiology; Dental implants; Overdenture
MeSH Terms: conditions — Nutrition Disorders; Jaw, Edentulous

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study examines the effects of prosthetic treatment options applied to edentulous geriatric individuals who applied to Marmara University Faculty of Dentistry on chewing function, food consumption status, malnutrition status and oral health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 50 years old,
* Those who volunteer to participate in the study,
* Those who have adequate bone height and thickness in the intraforaminal region
* Those who have Upper and lower fully edentulous jaws

Exclusion Criteria:

* Those who have systemic diseases that may cause systemic neuropathy, such as diabetes, hypertension, kidney disease,
* Those who do not want to sign the consent form,
* Clinical or radiographic pathological condition in the intraforaminal region
* Patients with a history of malignancy, radiotherapy or chemotherapy will be excluded from the study.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients over 50, who were admitted to Marmara University Faculty of Dentistry, Department of Oral and Maxillofacial Surgery, to have two implant-supported overdenture prostheses made, will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Change in chewing ability | 9 months
  In this study, a questionnaire consisting of open and closed-ended questions will be used to determine the chewing difficulties of individuals. With open-ended questions, foods that are difficult to chew and the methods used to consume these foods will be questioned. In the follow-up interviews, closed-ended questions such as the ability to chew the previously listed foods are "easy to chew", "I have a little difficulty", "I have a lot of difficulty / can't chew at all". If individuals say, "I have a little or a lot of difficulty" while chewing hard foods and "I have some or a lot of difficulty" when chewing soft foods, they will be evaluated as "difficulty in chewing". At baseline, 3 months after temporary complete denture treatment, 3 and 6 months after implant-supported overdenture treatment, the chewing ability will be determined.
Change in Malnutrition Status | 9 months
  The Mini Nutritional Assessment (MNA) will be used to assess changes in nutritional status. MNA is an easy-to-apply, low-cost and reliable method that is frequently used in the evaluation of malnutrition status. The MNA consists of 4 parts. These four parts; anthropometric assessment (BMI, weight, arm and calf circumferences); general status assessment (lifestyle, medication, mobility, cognition/depression); short nutritional assessment (number of full meals, food and liquids intake, self-sufficiency in eating) and subjective assessment (self-perception about health and nutrition status). MNA classifies elderly patients as good status (scores ≥ 24), risk of malnutrition (scores between 17-23.5), or malnourished (scores <17). MNA will be applied by the researchers in face-to-face meetings within baseline, 3 months after temporary complete denture treatment, 3 and 6 months after implant-supported overdenture treatment
Change in food consumption | 9 months
  To evaluate the food consumption of the geriatric individuals included in the study, at baseline, 3 months after temporary complete denture treatment, 3 and 6 months after implant-supported overdenture treatment will be taken with 24-hour recall method. The amount of nutrients included in the meals will be calculated by using the "Standard Recipes" book, and the measurement amounts will be calculated by using the "Food Photo Catalogue" book. The data obtained from the 24-hour recall method will be analyzed using the "Computer Assisted Nutrition Program, Nutrition Information Systems Package Program (BEBIS)" and the amount of energy, carbohydrates, protein, fat, fiber and micronutrients consumed by participants will be calculated. Intake of energy, macro nutrients, fiber and micronutrients will be compared with the baseline, 3 months after temporary complete denture treatment, 3 and 6 months after implant-supported overdenture treatment.
Change in body composition | 9 months
  Body composition consists of body fluid, body fat, muscle mass and bone components. The sum of bone and muscle mass gives lean body mass. For body composition analysis, an 8-electrode bioelectrical impedance (BIA) device Tanita MC 780 MA, which performs segmental analysis, will be used. Individuals will be asked to remove all metal items (rings, earrings, bracelets, watches, phones, etc.), any heavy clothing, shoes, and socks before stepping on the device. The device is set to -1.0 kg for the remaining clothes. With this measurement, which takes about 1 minute, the body weight (kg), total body fluid (kg), total body fat (kg), lean body mass (kg) and muscle mass (kg) values will be obtained.

SECONDARY OUTCOMES:
Change in Oral-Health Impact Profile | 9 months
  A scale of 1 to 5 will be used to rate each of the 14 questions about how dental health affects quality of life (minimum score of 0, maximum score of 70). Higher ratings reflect a greater influence of the patient's dental health on their quality of life (higher scores, worse outcomes). At baseline, 3 months after temporary complete denture treatment, 3 and 6 months after implant-supported overdenture treatment, the questionnaire will be taken.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University School of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Akoglu B, Ucankale M, Ozkan Y, Kulak-Ozkan Y. Five-year treatment outcomes with three brands of implants supporting mandibular overdentures. Int J Oral Maxillofac Implants. 2011 Jan-Feb;26(1):188-94. PMID 21365055
- [Background] Cousson PY, Bessadet M, Nicolas E, Veyrune JL, Lesourd B, Lassauzay C. Nutritional status, dietary intake and oral quality of life in elderly complete denture wearers. Gerodontology. 2012 Jun;29(2):e685-92. doi: 10.1111/j.1741-2358.2011.00545.x. Epub 2011 Oct 17. PMID 22004061
- [Background] Kossioni A, Bellou O. Eating habits in older people in Greece: the role of age, dental status and chewing difficulties. Arch Gerontol Geriatr. 2011 Mar-Apr;52(2):197-201. doi: 10.1016/j.archger.2010.03.017. PMID 20399518
- [Background] Lamy M, Mojon P, Kalykakis G, Legrand R, Butz-Jorgensen E. Oral status and nutrition in the institutionalized elderly. J Dent. 1999 Aug;27(6):443-8. doi: 10.1016/s0300-5712(99)00002-0. PMID 10399411
- [Background] Sheiham A, Steele JG, Marcenes W, Lowe C, Finch S, Bates CJ, Prentice A, Walls AW. The relationship among dental status, nutrient intake, and nutritional status in older people. J Dent Res. 2001 Feb;80(2):408-13. doi: 10.1177/00220345010800020201. PMID 11332523
- [Background] Slade GD, Spencer AJ. Development and evaluation of the Oral Health Impact Profile. Community Dent Health. 1994 Mar;11(1):3-11. PMID 8193981
- [Background] Slade GD. Derivation and validation of a short-form oral health impact profile. Community Dent Oral Epidemiol. 1997 Aug;25(4):284-90. doi: 10.1111/j.1600-0528.1997.tb00941.x. PMID 9332805
- [Background] Ucankale M, Akoglu B, Ozkan Y, Ozkan YK. The effect of different attachment systems with implant-retained overdentures on maximum bite force and EMG. Gerodontology. 2012 Mar;29(1):24-9. doi: 10.1111/j.1741-2358.2010.00389.x. Epub 2010 Jun 30. PMID 20604812